CLINICAL TRIAL: NCT01733004
Title: A Phase 1 Study of MM-141 in Patients With Advanced Solid Tumors
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Merrimack Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: MM-141-01-01-01
Record Dates: First submitted 2012-11-20; First posted 2012-11-26 (Estimated); Last update posted 2016-08-04 (Estimated); Status verified 2016-08

CONDITIONS: Hepatocellular Carcinoma
Keywords: Cancer; Hepatocellular Carcinoma; Oncology; Phase I; ErbB3; IGF-1R; Everolimus; Gemcitabine; Abraxane
MeSH Terms: conditions — Carcinoma, Hepatocellular; Neoplasms; Insulin-Like Growth Factor I, Resistance To | interventions — Istiratumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Arm A (Experimental): MM-141 monotherapy
  Interventions: Drug: MM-141
- Arm B (Experimental): MM-141 and Everolimus
  Interventions: Drug: MM-141
- Arm C (Experimental): MM-141 and Abraxane and Gemcitabine
  Interventions: Drug: MM-141

INTERVENTIONS:
Drug: MM-141

SUMMARY:
This study is a Phase 1 and pharmacologic open-labeled dose-escalation trial using a "3+3" design, evaluating MM-141 at varying dose levels and frequencies.

ELIGIBILITY:
Inclusion Criteria:

* Advanced malignant solid tumors for which no curative therapy exists that has recurred or pgrogressed following standard therapy
* Eighteen years of age or above
* Able to understand and sign an informed consent (or have a legal representative who is able to do so)
* Measurable disease according to RECIST v1.1
* ECOG Performance Score of 0 or 1
* Adequate bone marrow, hepatic, renal and cardiac function
* Willing to abstain from sexual intercourse or to use an effective form of contraception during the study and for 90 days following the last dose of MM-141

Exclusion Criteria:

* Active infection or fever > 38.5°C during screening visits or on the first scheduled day of dosing
* Symptomatic CNS disease
* Received other recent antitumor therapy
* Pregnant or breast feeding

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 42 (Actual)
Dates: Start 2012-11; Primary Completion 2016-01 (Actual)

PRIMARY OUTCOMES:
Severity and number of adverse events related to escalating doses of MM-141 | 2 years
  Determine the Phase II dose based either on the maximum tolerated dose (MTD) or recommended dose in patients with advanced solid malignancies.

CONTACTS AND LOCATIONS:
Overall Officials: Chrystal Louis, MD, MPH, Study Director — Merrimack Pharmaceuticals
Locations (4):
- United States (3):
  - Marietta, Georgia
  - Boston, Massachusetts
  - Detroit, Michigan
- Villejuif, France